CLINICAL TRIAL: NCT06807229
Title: Core Stability vs. Traditional Physical Therapy: A Comparative Study on Alleviating Low Back Pain in Dysmenorrhea
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Middle East University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AhmedM
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Dysmenorrhea; Low Back Pain
Keywords: Dysmenorrhea; Low back pain; core stability
MeSH Terms: conditions — Dysmenorrhea; Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: A convenient sample of 80 participants will be screened for study eligibility. The sample size was calculated utilizing G*Power based on a prior study with an effect size of 0.8. to detect a true difference in means with 80% power and a 5% significance level. An estimated sample size of 70 patients will be randomly allocated to a software application.
  Group A will receive core stability exercises combined traditional physical therapy (stretching exercises and TENS). The 2nd group (group B) will receive traditional physical therapy (stretching exercises and TENS) only.
  Randomization Informed consent will be attained from each individual after explanation of the aim as well as benefits of the study. Individuals were informed about the privacy of their information and their right to stop or withdraw at any time. They will be randomized using the randomization block method into two groups, study (n=35) and control (n=35) groups.
Who Masked: Participant
Masking Description: A convenient sample of 80 participants will be screened for study eligibility. The sample size was calculated utilizing G*Power based on a prior study with an effect size of 0.8. to detect a true difference in means with 80% power and a 5% significance level. An estimated sample size of 70 patients will be randomly allocated to a software application. Group A will receive core stability exercises combined traditional physical therapy (stretching exercises and TENS). The 2nd group (group B) will receive traditional physical therapy (stretching exercises and TENS) only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- core stability exercise group (Experimental): Subjects in this group will be handled with core stability exercises that targeted deep abdominal muscles. This included a series of exercises as well as a baseline therapeutic management of ultrasonic as well as TENS. A physiotherapist supervised these exercises.
  For four weeks, all groups did core stability exercises for 30 minutes three times per week. Isometric contraction was sustained for 7-8 seconds for every exercise. Each exercise was repeated ten times, with a three-second rest break among repetitions. Patients were given a 1-minute break between exercises. (13) Based on the patient's success, the intensity of the individual training steadily increased with decreasing therapist support. Patients were told to contract their abdominal muscles and hold the contraction while continuing to breathe normally during each repetition of each exercise. (22) Each patient followed a customized exercise program designed by their therapist and kept track of their progress in a diary.
  Interventions: Device: Transcutaneous electrical nerve stimulation; Other: stretching exercises
- traditional physical therapy (Active Comparator): Stretching exercises Information will be given to participants of group (A) to do 4 stretching exercises for 8 weeks at home (3 days per week and 3 times per day for 10 minutes). They were asked to avoid performing stretching exercises during the period cycle. They will be given a questionnaire prior to the stretching exercises and completed it after 4 weeks of stretching exercises Transcutaneous electrical nerve stimulation (TENS) We will apply high frequency TENS for low back pain relief as it showed effectiveness more than low frequency TENS in pain relief (21). The recommendation is to apply the TENS at the highest tolerable intensity (22). While adjusting the current amplitude in a continuous manner so that its presence will be noticeable throughout the treatment. We applied a TENS device (ENRAF NONIUS Model, four electrodes) with a frequency of 0- 100/HZ and 90-100 pulse /seconds was applied for 20 minutes, to increase circulation and to have pain relief
  Interventions: Device: Transcutaneous electrical nerve stimulation; Other: stretching exercises

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — We will apply high frequency TENS for low back pain relief as it showed effectiveness more than low frequency TENS in pain relief (21). The recommendation is to apply the TENS at the highest tolerable intensity (22). While adjusting the current amplitude in a continuous manner so that its presence will be noticeable throughout the treatment. We applied a TENS device (ENRAF NONIUS Model, four electrodes) with a frequency of 0- 100/HZ and 90-100 pulse /seconds was applied for 20 minutes, to increase circulation and to have pain relief at the first day of menstrual complaints without taking any analgesics. Patients lied in prone position with a thin pillow placed under their abdomen. Two electrodes were placed to the proximal margin of low back area, and two others were placed to the proximal of gluteal region laterally. The intensity of stimulation was increased up to the tolerated level without causing any contraction
  Other Names: TENS; stretching exercises
Other: stretching exercises — The first stretching exercise: The subjects will be asked to stand and bend trunk forward from the hip joint so that the shoulders and back were positioned on a straight line and the upper body was placed parallel to the floor for 5 seconds repetition; 10 times.
  The second stretching exercise: The subjects will be requested to stand then raise 1 heel off the floor, then repeat the exercise with the other heel alternatively. The exercise will be performed 20 times.
  The third stretching exercise: The subjects will be asked to spread their feet shoulder width, place trunk and hands in forward stretching.
  The fourth stretching exercise: The subjects will be asked to spread her feet wider than shoulder width. Then the subject was asked to bend and touch left ankle with her right hand while putting her left hand in a stretched position above her head so that the head was in the middle and her head was turned and looked for her left hand, this exercise was repeated for the opposite foot with
  Other Names: TENS

SUMMARY:
Dysmenorrhea is a menstrual disorder defined by the presence of painful cramps of uterine origin that occur during menstruation. It is one of the most common causes of pelvic pain and short-term absenteeism from school or work, among young and adult women [1].

The prevalence of Primary dysmenorrhea is highest in the 16-25-year age group but is greatly underestimated as many women consider pain a normal part of the menstrual cycle and do not seek medical treatment, despite the considerable distress they experience. A previous systematic review on the impact of dysmenorrhea in adolescents reported that the prevalence is high and that it imposes a significant negative impact on academic performance [2], restrictions on daily activities and sports or social and sexual relationships [3].

Primary dysmenorrhea occurs in the absence of pelvic pathology, it is mediated by elevated prostaglandin and leukotriene levels, inflammation causing uterine contractility and cramping pain. Secondary dysmenorrhea is due to pelvic pathology or a recognized medical condition and accounts for about 10% of cases of dysmenorrhea. The most common etiology of secondary dysmenorrhea is endometriosis, other etiologies include congenital or acquired obstructive and nonobstructive anatomic abnormalities (e.g., müllerian malformations, uterine leiomyomas, adenomyosis), pelvic masses, and infection [4].

It has been demonstrated that prostaglandins are overproduced in dysmenorrhea. Prostaglandins cause narrowing of the blood vessels supplying the uterus, abnormal contractile activity of the uterus, which leads to ischemia, hypoxia of the uterus and increased sensitivity of the nerve endings [5].

The treatment approach is mainly directed toward relieving the pain through physiological mechanisms that underlie menstrual pain (production of prostaglandins). The treatment is also aimed toward the improvement of the function, leading to fewer days lost at work, school or extracurricular activities [6]. There are different approaches to the treatment of primary dysmenorrhea. The drug approach is achieved through prostaglandins inhibitors, which are non-steroidal anti-inflammatory drugs (NSAIDs) and hormonal drugs such as contraceptives. Many NSAIDs which non-specifically inhibit both COX-1 and COX-2 enzymes (e.g., ibuprofen) are the most common initial therapy for dysmenorrhea [7]. Likewise, oral contraceptives are not free from side effects either, related as they are to the frequency of bleeding, weight gain, or the patient's basal risk of venous thromboembolism [1].

All this shows us that there is a need for emphasis on alternative methods of conservative treatment as a non-pharmacological and non-invasive therapy, safe and easy to use for obtaining relief from dysmenorrhea symptoms, including acupuncture and acupressure, biofeedback, heat treatments, transcutaneous electrical nerve stimulation (TENS), exercises and relaxation techniques [8]. On the other hand, these physiotherapeutic treatments, being supported by clinical trial data, could be a very useful treatment alternative for women with primary dysmenorrhea, particularly those who are not eligible for pharmacological therapy, since physiotherapy has no side effects according to the analyzed studies [9]. Exercise is an activity performed to develop or maintain fitness which requires physical exertion, is one of the non-pharmacological and effective ways of treating dysmenorrhea. Many reviews have evaluated the efficacy of exercise or individual physiotherapy interventions for primary dysmenorrhea [10].

Alternative or non-pharmacological treatments include TENS, exercise, acupuncture, acupressure, massage therapy, heat pads. The reduction of pain maybe due to the effect's hormonal changes in the uterine tissue or due to an increase in the endorphin levels [11].

Core muscle strengthening focuses on isolated muscle group conditioning which will strengthen the small intrinsic musculature around the lumbar spine and provide lumbar stability. When these muscles are strong, they become capable of handling normal biomechanical forces even the stress of menstrual cramps which a women's body undergoes during the menstrual cycle (12).

Core stability exercise has been known as a beneficial intervention in the management of several medical problems. Core stability exercises strengthen and coordinate the muscles around the abdominal, lumbar, and pelvic regions. Because it has been suggested that the core stability exercises mainly affect the lumbosacral muscles and increase blood supply in lumbosacral structures.

It was proved in some studies that core stability exercises can improve pain and function for primary dysmenorrhea in young and adult women. (13,14) but the number of studies about this were limited with many limitations so, we hypothesized that the core stability exercises might be effective in reducing primary dysmenorrhea symptoms.

So, this study was designed to compare among the effect

DETAILED DESCRIPTION:
Core Stability vs. Traditional Therapy: A Comparative Study on Alleviating Low Back Pain in Dysmenorrhea Dysmenorrhea is a menstrual disorder defined by the presence of painful cramps of uterine origin that occur during menstruation. It is one of the most common causes of pelvic pain and short-term absenteeism from school or work, among young and adult women [1].

The prevalence of Primary dysmenorrhea is highest in the 16-25-year age group but is greatly underestimated as many women consider pain a normal part of the menstrual cycle and do not seek medical treatment, despite the considerable distress they experience. A previous systematic review on the impact of dysmenorrhea in adolescents reported that the prevalence is high and that it imposes a significant negative impact on academic performance [2], restrictions on daily activities and sports or social and sexual relationships [3].

Primary dysmenorrhea occurs in the absence of pelvic pathology, it is mediated by elevated prostaglandin and leukotriene levels, inflammation causing uterine contractility and cramping pain. Secondary dysmenorrhea is due to pelvic pathology or a recognized medical condition and accounts for about 10% of cases of dysmenorrhea. The most common etiology of secondary dysmenorrhea is endometriosis, other etiologies include congenital or acquired obstructive and nonobstructive anatomic abnormalities (e.g., müllerian malformations, uterine leiomyomas, adenomyosis), pelvic masses, and infection [4].

It has been demonstrated that prostaglandins are overproduced in dysmenorrhea. Prostaglandins cause narrowing of the blood vessels supplying the uterus, abnormal contractile activity of the uterus, which leads to ischemia, hypoxia of the uterus and increased sensitivity of the nerve endings [5].

The treatment approach is mainly directed toward relieving the pain through physiological mechanisms that underlie menstrual pain (production of prostaglandins). The treatment is also aimed toward the improvement of the function, leading to fewer days lost at work, school or extracurricular activities [6]. There are different approaches to the treatment of primary dysmenorrhea. The drug approach is achieved through prostaglandins inhibitors, which are non-steroidal anti-inflammatory drugs (NSAIDs) and hormonal drugs such as contraceptives. Many NSAIDs which non-specifically inhibit both COX-1 and COX-2 enzymes (e.g., ibuprofen) are the most common initial therapy for dysmenorrhea [7]. Likewise, oral contraceptives are not free from side effects either, related as they are to the frequency of bleeding, weight gain, or the patient's basal risk of venous thromboembolism [1].

All this shows us that there is a need for emphasis on alternative methods of conservative treatment as a non-pharmacological and non-invasive therapy, safe and easy to use for obtaining relief from dysmenorrhea symptoms, including acupuncture and acupressure, biofeedback, heat treatments, transcutaneous electrical nerve stimulation (TENS), exercises and relaxation techniques [8]. On the other hand, these physiotherapeutic treatments, being supported by clinical trial data, could be a very useful treatment alternative for women with primary dysmenorrhea, particularly those who are not eligible for pharmacological therapy, since physiotherapy has no side effects according to the analyzed studies [9]. Exercise is an activity performed to develop or maintain fitness which requires physical exertion, is one of the non-pharmacological and effective ways of treating dysmenorrhea. Many reviews have evaluated the efficacy of exercise or individual physiotherapy interventions for primary dysmenorrhea [10].

Alternative or non-pharmacological treatments include TENS, exercise, acupuncture, acupressure, massage therapy, heat pads. The reduction of pain maybe due to the effect's hormonal changes in the uterine tissue or due to an increase in the endorphin levels [11].

Core muscle strengthening focuses on isolated muscle group conditioning which will strengthen the small intrinsic musculature around the lumbar spine and provide lumbar stability. When these muscles are strong, they become capable of handling normal biomechanical forces even the stress of menstrual cramps which a women's body undergoes during the menstrual cycle (12).

Core stability exercise has been known as a beneficial intervention in the management of several medical problems. Core stability exercises strengthen and coordinate the muscles around the abdominal, lumbar, and pelvic regions. Because it has been suggested that the core stability exercises mainly affect the lumbosacral muscles and increase blood supply in lumbosacral structures.

It was proved in some studies that core stability exercises can improve pain and function for primary dysmenorrhea in young and adult women. (13,14) but the number of studies about this were limited with many limitations so, we hypothesized that the core stability exercises might be effective in reducing primary dysmenorrhea symptoms.

So, this study was designed to compare among the effect of core stability in relation to traditional treatment of primary dysmenorrhea.

Subjects and methods This study is a randomized controlled study. All procedures used in the study will be compliant with the Declaration of Helsinki, which regulates research involving human subjects. Registration Clinical Trial Registration database (?) and approval from the Faculty of Physical Therapy, Delta University's institutional review board (No: ?). This study was carried out at outpatient clinic at faculty of physical therapy, delta university for science and technology, Egypt. The registration and recruitment of individuals and follow-up procedures were done from November 2024 to March 2025.

Subjects:

The patients will be included in this study had these criteria: Females diagnosed with primary dysmenorrhea between age group 18-35 years and their VAS Score is 4 ≥, regular menstrual cycle, unmarried females, non-athlete.

The exclusion criteria: history of pelvic inflammatory disease, endometriosis, any pathology, compulsory use of special drugs, had symptoms such as (tingling, itching, discharge), Irregular menstruation cycle, use of painkillers during the study period, any musculoskeletal problems causing inability to perform core strengthening exercises, mental, psychological problems.

Sample size A convenient sample of 80 participants will be screened for study eligibility. The sample size was calculated utilizing G*Power based on a prior study with an effect size of 0.8. to detect a true difference in means with 80% power and a 5% significance level. An estimated sample size of 70 patients will be randomly allocated to a software application. Group A will receive core stability exercises combined traditional physical therapy (stretching exercises and TENS). The 2nd group (group B) will receive traditional physical therapy (stretching exercises and TENS) only.

Randomization Informed consent will be attained from each individual after explanation of the aim as well as benefits of the study. Individuals were informed about the privacy of their information and their right to stop or withdraw at any time. They will be randomized using the randomization block method into two groups, study (n=35) and control (n=35) groups. Allocation sequence will be applied by a blinded and independent research assistant who opened sealed envelopes containing a computer-generated randomized number.

Assessment procedures:

The assessors who participated in this study will be blinded to the patients' allocation in the studied groups. The outcome measures of this study were evaluated by one physiotherapist with an experience of more than 10 years in musculoskeletal and neurological conditions. Evaluating the pain severity & functional quality of life and core stability measures were conducted for all patients before commencing the treatment and immediately after completing the treatment period of 4 weeks in the following order:

1. Pain severity for lumbar region:

   We will use Visual Analogue Scale (VAS) which is a reliable and effective tool of pain intensity that is sensitive to variations in pain caused by clinical conditions, was used to assess the severity of the pain. At the scale's left end, a zero means there is no pain, and a 10 means the most agonizing suffering possible. A minor improvement with a change of 1.1-1.2 cm is clinically meaningful. (15)
2. Arabic oswestry disability index AODI assessment:

   Patients will complete a questionnaire, which indicates a percentage score of level of function in daily living activities in pre-sessions and after end of sessions. This questionnaire examines levels of function every day in ten daily living activities. The categories will be scored from zero to five (10 categories). If all 10 sectors are finished the result is calculated as follows: if 20 the total result out of 50 total possible, score x 100 = 40%. (14) We recorded the results of this scale before and after the study. (15)
3. WaLIDD score:

   It is a scale-type survey and abbreviation of (working ability, location, intensity, days of pain, dysmenorrhea), score: 0 without dysmenorrhea, 1-4 mild dysmenorrhea, 5-7 moderate dysmenorrhea, 8-12 severe dysmenorrhea. Wong-Baker scale was reclassified to adjust a four-level scale. We recorded the results of this scale before and after the study. (18) We will record the results of this scale before and after the study.
4. Core stability endurance test:

They are three core endurance tests generated by McGgill. (19) they are trunk flexor test, trunk extensor test and side bridge test. The trunk flexor test was performed while the body was 60° in flexion, knees and hip were 90° in flexion. The arms were joined diagonally on the chest. Participants were wanted to protect this position as long as it is possible. The test was terminated when the individual could not maintain this position. The trunk extensor test was performed on the treatment table in a prone position. Pelvis, hip and knees were fixed to the treatment table up to spina iliaca anterior superior level. The body and upper extremities were supported with a chair at the same height as the surface of the table. Then the chair was removed and the individual tried to keep the horizontal body position as long as possible while crossing the arms on the chest. The test was terminated when the person fell below the horizontal position. The side bridge test was performed on the dominant side on the mat. Because no difference between the left and right side has been previously reported, only the dominant side was evaluated (12). Knees of the participants were on the extensions with same line of feet. Body weight was supported only by the lower elbows and feet while lifting her hips on the mat. The test was terminated when the side-lying position deteriorated and the hip fell. The measurement results of McGill endurance test recorded in seconds.

Intervention procedures:

Core stability exercises (CSE): Subjects in this group will be handled with core stability exercises that targeted deep abdominal muscles. This included a series of exercises as well as a baseline therapeutic management of ultrasonic as well as TENS. A physiotherapist supervised these exercises.

For four weeks, all groups did core stability exercises for 30 minutes three times per week. Isometric contraction was sustained for 7-8 seconds for every exercise. Each exercise was repeated ten times, with a three-second rest break among repetitions. Patients were given a 1-minute break between exercises. (13) Based on the patient's success, the intensity of the individual training steadily increased with decreasing therapist support. Patients were told to contract their abdominal muscles and hold the contraction while continuing to breathe normally during each repetition of each exercise. (22) Each patient followed a customized exercise program designed by their therapist and kept track of their progress in a diary. The core stabilization exercises included the abdominal hollowing, supine extension bridging, straight leg raising from prone. As shown in (Table 1), various CSE methods have been developed.

TABLE 1. Details of the core stabilization exercises Type of Exercise Description abdominal hollowing The therapist was standing at the patient's waist, and she spread her fingers laterally toward the rectus abdominis muscles and positioned her thumbs anteriorly and inferiorly to the ASIS. The patient took the usual laying posture. The next step was to have the patient contract her abdominal muscles and hold a downward pressure on her lower back. (figure 2) Supine extension bridge Both of the participant's feet are placed below the knees in a hook-lying position. By gradually rising his or her hips until his or her knees as well as shoulders are aligned in a straight line, the individual shifts the body's weight to the shoulders instead of the neck. After holding this position, the individual slowly drops his or her hips to the floor. (figure 3a & b) Straight leg rise from prone The participant lies on his or her back with their heads resting on their arms. The participant elevates his or her right leg as high as they can toward the ceiling by contracting the gluteus and hamstring muscles in that leg. The participant holds this still position before gradually lowering one leg. Repeat the drill on the left side. (figure 4a & b)

Traditional Physiotherapy program Stretching exercises

Information will be given to participants of group (A) to do 4 stretching exercises for 8 weeks at home (3 days per week and 3 times per day for 10 minutes). They were asked to avoid performing stretching exercises during the period cycle. They will be given a questionnaire prior to the stretching exercises and completed it after 4 weeks of stretching exercises (10). The prescribed exercises were as follows:

The first stretching exercise: The subjects will be asked to stand and bend trunk forward from the hip joint so that the shoulders and back were positioned on a straight line and the upper body was placed parallel to the floor for 5 seconds repetition; 10 times.

The second stretching exercise: The subjects will be requested to stand then raise 1 heel off the floor, then repeat the exercise with the other heel alternatively. The exercise will be performed 20 times.

The third stretching exercise: The subjects will be asked to spread their feet shoulder width, place trunk and hands in forward stretching.

The fourth stretching exercise: The subjects will be asked to spread her feet wider than shoulder width. Then the subject was asked to bend and touch left ankle with her right hand while putting her left hand in a stretched position above her head so that the head was in the middle and her head was turned and looked for her left hand, this exercise was repeated for the opposite foot with the same method. The exercises were repeated alternatively 10 times for each side of the body

Transcutaneous electrical nerve stimulation (TENS) We will apply high frequency TENS for low back pain relief as it showed effectiveness more than low frequency TENS in pain relief (21). The recommendation is to apply the TENS at the highest tolerable intensity (22). While adjusting the current amplitude in a continuous manner so that its presence will be noticeable throughout the treatment. We applied a TENS device (ENRAF NONIUS Model, four electrodes) with a frequency of 0- 100/HZ and 90-100 pulse /seconds was applied for 20 minutes, to increase circulation and to have pain relief at the first day of menstrual complaints without taking any analgesics. Patients lied in prone position with a thin pillow placed under their abdomen. Two electrodes were placed to the proximal margin of low back area, and two others were placed to the proximal of gluteal region laterally. The intensity of stimulation was increased up to the tolerated level without causing any contraction (23)

Reference

1. Bernardi, M., Lazzeri, L., Perelli, F., Reis, F.M., Petraglia, F. 2107: "Dysmenorrhea and related disorders". F1000Research (6): 1645.
2. Armour, M., Parry, K., Manohar, N., Holmes, K., Ferfolja, T., Curry, C. 2019: "The Prevalence and Academic Impact of Dysmenorrhea in 21,573 Young Women: A Systematic Review and Meta-Analysis" J. Women's Health: (28): 1161-1171.
3. Orhan, C., Celenay, S.T., Demirtuerk, F., Ozgul, S., Uzelpasaci, E., Akbayrak, T. 2018: " Effects of menstrual pain on the academic performance and participation in sports and social activities in Turkish university students with primary dysmenorrhea: A case control study. J. Obstet. Gynaecol" Res. ( 44): 2101-2109.
4. ACOG committee opinion no. 760. 2018: "dysmenorrhea and endometriosis in the adolescent" Obstet. Gynecol. 132(6): 249-258.
5. Barcikowska, Z., Rajkowska-Labon, E., Grzybowska, M.E., Hansdorfer-Korzon, R., Zorena, K. 2020: " Inflammatory markers in dysmen orrhea and therapeutic options. Int. J. Environ" Res. Public Health. (17):1191.
6. Ryan, S.A. 2019: " The Treatment of Dysmenorrhea" Pediatr. Clin. N. Am. (64): 331-342.
7. Yacubovich, Y., Cohen, N., Tene, L., Kalichman, L. 2019: "The prevalence of primary dysmenorrhea among students and its association with musculoskeletal and myofascial pain". J. Bodyw. Mov. Ther. (23): 785-791.
8. Fernández-Martínez, E., Onieva-Zafra, M.D., Parra-Fernández, M.L. 2019: "The impact of dysmenorrhea on quality of life among spanish female university students" Int. J. Environ. Res. Public Health. (16): 713.
9. Arik, M.I., Kiloatar, H., Aslan, B., Icelli, M. 2020: "The effect of tens for pain relief in women with primary dysmenorrhea: A systematic review and meta-analysis. Explore. (29): 2541.
10. Saleh HS, Mowafy HE, El Hameid A. 2016: "Stretching or core strengthening exercises for managing primary dys menorrhea". J Women's Health Care. 5(295): 2167-0420.
11. Shahrjerdi, Shahnaz, et al. "Effect of core stability exercises on primary dysmenorrhea: a randomized controlled trial." Journal of Modern Rehabilitation 13.2 (2019): 113-122.
12. Zainab, S., et al. "A study to compare the effectiveness of core strengthening exercises for phase I and phase II of menstrual cycle in primary dysmenorrhea subjects." Biomedicine 41.2 (2021): 315-317.
13. Shahnaz S., Fahimeh M., Rahman S. and Samira S. 2019: " Effect of Core Stability Exercises on Primary Dysmenorrhea: A Randomized Controlled Trial". Journal of Modern Rehabilitation. 13(1):113-122.
14. Shafshak TS, Elnemr R. The Visual Analogue Scale Versus Numerical Rating Scale in Measuring Pain Severity and Predicting Disability in Low Back Pain. J Clin Rheumatol. 2021 Oct 1;27(7):282-285.
15. Algarni A, Ghorbel S, Jones J et al. (2014): Validation of an Arabic version of the Oswestry index in Saudi Arabia. Annals of Physical and Rehabilitation Medicine, 57 (9-10): 653-63.
16. Teherán AA, Piñeros LG, Pulido F, Mejía Guatibonza MC. WaLIDD score, a new tool to diagnose dysmenorrhea and predict medical leave in university students. International journal of women's health. 2018 Jan 17:35-45.
17. McGill, S. (2006). Ultimate back fitness and performance (pp. 277-285). Backfitpro Incorporated.
18. Kanik ZH, Pala OO, Gunaydin G, et al. Relationship between scapular muscle and core endurance in healthy subjects. J Back Musculoskelet Rehabil 2017;30:811-17.
19. Saleh MSM, Botla AMM, Elbehary NAM. Effect of core stability exercises on postpartum lumbopelvic pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(2):205-213.
20. Roostayi MM (2000) Physiotherapy and exercise therapy in women and obstetric. Sana Nashr, Tehran.
21. Lauretti GR, Oliveira R, Parada F, Mattos AL. The new portable transcutaneous electrical nerve stimulation device was efficacious in the control of primary dysmenorrhea cramp pain. Neuromodulation. 2015;18(6):522-527. doi:10.1111/ner.12269
22. Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014;4(3):197-209. doi:10.2217/pmt.14.13
23. Parsa, Parisa, and Saeed Bashirian. "Effect of transcutaneous electrical nerve stimulation (TENS) on primary dysmenorrhea in adolescent girls." Journal of Postgraduate Medical Institute 27.3 (2013).

ELIGIBILITY:
Inclusion Criteria: Females diagnosed with primary dysmenorrhea between age group 18-35 years and their VAS Score is 4 ≥, regular menstrual cycle, unmarried females, non-athlete.

Exclusion Criteria: history of pelvic inflammatory disease, endometriosis, any pathology, compulsory use of special drugs, had symptoms such as (tingling, itching, discharge), Irregular menstruation cycle, use of painkillers during the study period, any musculoskeletal problems causing inability to perform core strengthening exercises, mental, psychological problems

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females diagnosed with primary dysmenorrhea between age group 18-35 years and their VAS Score is 4 ≥, regular menstrual cycle, unmarried females, non-athlete.
Enrollment: 70 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | pre the intervention and immediately after the intervention
  The Visual Analogue Scale (VAS), a reliable and effective measure of pain intensity that is sensitive to variations in pain caused by clinical conditions, was used to assess the severity of the pain. At the scale's left end, a zero means there is no pain, and a 10 means the most agonizing suffering possible. A minor improvement with a change of 1.1-1.2 cm is clinically meaningful.
Arabic oswestry disability index AODI assessment | pre the intervention and immediately after the intervention
  Patients will complete a questionnaire, which indicates a percentage score of level of function in daily living activities in pre-sessions and after end of sessions. This questionnaire examines levels of function every day in ten daily living activities. The categories will be scored from zero to five (10 categories). If all 10 sectors are finished the result is calculated as follows: if 20 the total result out of 50 total possible, score x 100 = 40%. (14) We recorded the results of this scale before and after the study
WaLIDD score | pre the intervention and immediately after the intervention
  It is a scale-type survey and abbreviation of (working ability, location, intensity, days of pain, dysmenorrhea), score: 0 without dysmenorrhea, 1-4 mild dysmenorrhea, 5-7 moderate dysmenorrhea, 8-12 severe dysmenorrhea. Wong-Baker scale was reclassified to adjust a four-level scale. We recorded the results of this scale before and after the study
Core stability endurance test | pre the intervention and immediately after the intervention
  They are three core endurance tests generated by McGgill. (19) they are trunk flexor test, trunk extensor test and side bridge test. The trunk flexor test was performed while the body was 60° in flexion, knees and hip were 90° in flexion. The arms were joined diagonally on the chest. Participants were wanted to protect this position as long as it is possible. The test was terminated when the individual could not maintain this position. The trunk extensor test was performed on the treatment table in a prone position. Pelvis, hip and knees were fixed to the treatment table up to spina iliaca anterior superior level. The body and upper extremities were supported with a chair at the same height as the surface of the table. Then the chair was removed and the individual tried to keep the horizontal body position as long as possible while crossing the arms on the chest.

OTHER OUTCOMES:
age | pre the intervention only
  document the patient age through personal history information
weight | pre the intervention only
  we use weighing scale to measure weight of the subject in kilograms
height | pre the intervention only
  we measure height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- delta university for science and technology, Al Manşūrah, gamasah 11152, Gamasah, Al Manşūrah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided